CLINICAL TRIAL: NCT01346436
Title: Randomized Double Blind Controlled Trial of the Value of Robotic Rectopexy for the Treatment of Complex Pelvic Floor Dysfunction
Brief Title: Value of Robotic Rectopexy for the Treatment of Complex Pelvic Floor Dysfunction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nicolas C. Buchs (Other)
Responsible Party: Sponsor-Investigator, Nicolas C. Buchs, Faculty surgeon, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CER-11-047
Record Dates: First submitted 2011-04-29; First posted 2011-05-03 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Rectal Prolapse; Pelvic Organ Prolapse
MeSH Terms: conditions — Rectal Prolapse; Pelvic Organ Prolapse | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Robotic (Active Comparator): Use of daVinci surgical system (Intuitive Surgical Inc, Sunnyvale, CA) for the treatment of complex pelvic floor dysfunction
  Interventions: Procedure: Minimally invasive rectopexy
- Laparoscopy (Active Comparator): Use of standard laparoscopy for the treatment of complex pelvic floor dysfunction
  Interventions: Procedure: Minimally invasive rectopexy

INTERVENTIONS:
Procedure: Minimally invasive rectopexy — Use of a minimally invasive approach (robotic or laparoscopy) to perform a rectopexy
  Other Names: Surgery for rectal prolapse

SUMMARY:
The purpose of this randomized double blind controlled study is to assess the value of robotics for the treatment of complex pelvic floor dysfunction. The main aim is to compare perioperative and functional outcomes to the laparoscopic approach.

DETAILED DESCRIPTION:
Pelvic floor dysfunction is a common pathology. The management can be medical or surgical, depending on the location or the severity of the disease.

Since the large use of laparoscopy for the treatment of pelvic floor dysfunction, interesting and encouraging results have been published.

However, so far, a laparoscopic approach has some technical disadvantages like a poor ergonomy, a 2 dimensional vision, an unstable camera and the use of straight instruments. To overcome these natural limitations, robotics has been gaining increasing acceptance in general surgery.

Several groups have reported their encouraging experience with robotic rectopexy. Yet, these studies were not randomized or double blinded.

The aim of this study is to evaluate the role of robotics for complex pelvic floor dysfunction and to compare the outcomes to the laparoscopic approach.

ELIGIBILITY:
Inclusion Criteria:

* women
* proven pelvic floor dysfunction
* informed consent

Exclusion Criteria:

* Age <18 years old
* Patient unable to communicate or to understand the study
* Patient refusing to participate to the study
* contraindication to laparoscopy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-04; Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Perioperative outcomes | up to 30 days
  Including: blood loss, operative time, conversion rate, quality of dissection, pain, complications, hospital stay.

SECONDARY OUTCOMES:
Functional results | At 12 months
  Constipation score Incontinence score Quality of life score Sexuality score

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas C Buchs, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospital of Geneva, Department of Surgery, Geneva, Switzerland